CLINICAL TRIAL: NCT04401228
Title: Development and Validation of Predictive Models for Intensive Care Admission and Death of COVID-19 Patients in a Secondary Care Hospital in Belgium.
Brief Title: Predictive Models for Intensive Care Admission and Death of COVID-19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Clinique Saint Pierre Ottignies (Other)
Responsible Party: Principal Investigator, Nicolas Parisi, MD, Clinique Saint Pierre Ottignies
Other Study IDs: 0410508057
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: COVID19; Pneumonia, Viral; Inflammatory Response
Keywords: COVID19, prediction scores, ICU admission, death, TRIPOD.
MeSH Terms: conditions — COVID-19; Pneumonia, Viral; Death | interventions — Death Domain; Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- covid ICU patients
  Interventions: Other: predict admission of covid-19 patients to ICU and death with routine and quickly avalaible clinical, biological and radiological variables?
- covid conventionnal ward
  Interventions: Other: predict admission of covid-19 patients to ICU and death with routine and quickly avalaible clinical, biological and radiological variables?

INTERVENTIONS:
Other: predict admission of covid-19 patients to ICU and death with routine and quickly avalaible clinical, biological and radiological variables? — patients were questioned about their usual medication (Sartan, angiotensin-converting enzyme inhibitors, nonsteroidal anti-inflammatory drug, immunosuppressive drugs), their health condition (diabetes, hypertension, tobacco use, mental status). The Body mass index was computed.
  Age, gender, caucasian/african, weight, body mass index, number of days with symptoms before hospitalization, asthenia, pyrexia, dyspnea, chest pain, digestive sign, anosmia, ageusia, confusion, Travel or contact < one month, cigarette consumption ,hypertension, diabetes, mental status, angiotensin-converting-enzyme inhibitors, Sartan, non-steroidal anti-inflammatory drugs, immunosuppressive drugs, SpO2,Thoracic Computerized Tomography : % of lung injury, Thoracic Computerized Tomography : density of lung injury, blood type, white blood cells, neutrophils, lymphocytes, blood platelets, fibrinogen, ferritin, triglycerides, LDH, troponin, CRP. The dates of admission to ICU and death were recorded

SUMMARY:
To build simple and reliable predictive scores for intensive care admissions and deaths in COVID19 patients. These scores adhere to the TRIPOD (transparent reporting of a multivariable prediction model for individual prognosis or diagnosis) reporting guidelines.

The outcomes of the study are (i) admission in the Intensive Care Unit admission and (ii) death.

All patients admitted in the Emergency Department with a positive reverse transcription-polymerase chain reaction SARS-COV2 test were included in the study. Routine clinical and laboratory data were collected at their admission and during their stay. Chest X-Rays and CT-Scans were performed and analyzed by a senior radiologist.

Generalized Linear Models using a binomial distribution with a logit link function (R software version X) were used to develop predictive scores for (i) admission to ICU among emergency ward patients; (ii) death among ICU patients. A first panel of Number Models with the highest AIC (BIC) was preselected. Ten-fold cross-validation was then used to estimate the out-of-sample prediction error among these preselected models. The one with the smallest prediction error was in the end singled out .

ELIGIBILITY:
Inclusion Criteria:

* RT-PCR + SARS Cov2 pneumonia

Exclusion Criteria:

* < 18 ans -* GOLD 3 or 4 CPOD

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patient with COVID 19 with viral pneumonia
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
admission to ICU | through study completion, an average of 1 year

SECONDARY OUTCOMES:
death | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Saint-Pierre, Ottignies, Brabant Wallon, Belgium

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Rubin GD, Ryerson CJ, Haramati LB, Sverzellati N, Kanne JP, Raoof S, Schluger NW, Volpi A, Yim JJ, Martin IBK, Anderson DJ, Kong C, Altes T, Bush A, Desai SR, Goldin J, Goo JM, Humbert M, Inoue Y, Kauczor HU, Luo F, Mazzone PJ, Prokop M, Remy-Jardin M, Richeldi L, Schaefer-Prokop CM, Tomiyama N, Wells AU, Leung AN. The Role of Chest Imaging in Patient Management During the COVID-19 Pandemic: A Multinational Consensus Statement From the Fleischner Society. Chest. 2020 Jul;158(1):106-116. doi: 10.1016/j.chest.2020.04.003. Epub 2020 Apr 7. PMID 32275978
- [Background] Wynants L, Van Calster B, Collins GS, Riley RD, Heinze G, Schuit E, Bonten MMJ, Dahly DL, Damen JAA, Debray TPA, de Jong VMT, De Vos M, Dhiman P, Haller MC, Harhay MO, Henckaerts L, Heus P, Kammer M, Kreuzberger N, Lohmann A, Luijken K, Ma J, Martin GP, McLernon DJ, Andaur Navarro CL, Reitsma JB, Sergeant JC, Shi C, Skoetz N, Smits LJM, Snell KIE, Sperrin M, Spijker R, Steyerberg EW, Takada T, Tzoulaki I, van Kuijk SMJ, van Bussel B, van der Horst ICC, van Royen FS, Verbakel JY, Wallisch C, Wilkinson J, Wolff R, Hooft L, Moons KGM, van Smeden M. Prediction models for diagnosis and prognosis of covid-19: systematic review and critical appraisal. BMJ. 2020 Apr 7;369:m1328. doi: 10.1136/bmj.m1328. PMID 32265220
- [Background] Collins GS, Reitsma JB, Altman DG, Moons KG. Transparent Reporting of a multivariable prediction model for Individual Prognosis or Diagnosis (TRIPOD): the TRIPOD statement. Ann Intern Med. 2015 Jan 6;162(1):55-63. doi: 10.7326/M14-0697. PMID 25560714